CLINICAL TRIAL: NCT03826823
Title: Hysterosalpigography Using a Thin Catheter and Closing the Cervix With the Vaginal Speculum to Reduce the Pain
Brief Title: Thin Catheter for Hysterosalpigography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragaa Mansour, Director, The Egyptian IVF-ET Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-Mansour
Record Dates: First submitted 2011-07-11; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2008-03

CONDITIONS: Infertility
Keywords: hysterosalpingography, catheter, pain, visual analogue scale
MeSH Terms: conditions — Infertility; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- infertile women (Experimental): infertile women undergoing hysterosalpingography for evaluating fallopian tubes
  Interventions: Device: HSG cannula

INTERVENTIONS:
Device: HSG cannula — a thin catheter originally designed for IUI was introduced through the cervical canal into the lower part of the uterine cavity. After introducing the catheter, the screw of the vaginal speculum was loosened to allow the two valves of the speculum to press on the portiovaginalis of the cervix to prevent leakage of the dye. Then the dye was injected slowly and the procedure was watched on the screen and x-ray films were taken.

SUMMARY:
Hysterosalpingography is usually painful and the use of thin catheters of IUI could be an attractive alternative . we conducted a randomised controlled trial to compare the standard metal cannula to the thin catheter originally manufactured for intrauterine insemination. Pain assessment was done using visual analogue scale

DETAILED DESCRIPTION:
HSG is widely practiced in our country, however, for cost effective reasons, the standard metal cannula is the only method used at our hospital. It is painful procedure because it requires grasping the cervix with a tenaculum and inducing some cervical dilatation during introduction of the cannula. The aim of this pilot study was to modify the technique of HSG using a thinner than normal catheter, and without grasping the cervix with a tenaculum. Leakage of the dye through the cervix was prevented by pressing on the portiovaginalis of the cervix using the vaginal speculum.

ELIGIBILITY:
Inclusion Criteria:

* infertile women seeking evaluation of fallopian tubes

Exclusion Criteria:

* any woman with allergy to the iodine dye or condition contraindicating pregnancy

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
the level of pain using a visual analogue scale (VAS) | 8 month
  pain score will be assessed during introduction of catheter and during the injection of dye

SECONDARY OUTCOMES:
visualising uterus and tubes | 8 month
  the efficiency of the new technique in filling the uterine cavity with the dye and studying fallopian tubes.